CLINICAL TRIAL: NCT00757367
Title: A Phase 1, Open-Label, Controlled Clinical Trial to Determine the Pulmonary Residence Time of Insulin and Fumaryl Diketopiperazine, Utilizing Bronchoalveolar Lavage, After Administration of Technosphere® Insulin Inhalation Powder in Healthy Subjects
Brief Title: A Trial to Determine How Long Insulin and FDKP (the Molecule That Forms Technosphere Particles) Stays in the Lungs of Healthy Individuals After Inhalation of Technosphere® Insulin (TI) Powder Using Bronchoalveolar Lavage (BAL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-122
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Subjects
Keywords: Healthy subjects; insulin; bronchoscope; serum insulin; serum C-Peptide; BAL fluid; FDKP
MeSH Terms: conditions — Insulin Resistance

ARMS (1):
- TI Inhalation Powder (Experimental): TI Inhalation Powder, single dose, 60 units
  Interventions: Drug: TI Inhalation Powder

INTERVENTIONS:
Drug: TI Inhalation Powder — 1 60-U dose of TI Inhalation Powder before the bronchoscopy. Cohort 1 will undergo bronchoscopies at 30 minutes and again at 6 hours after the 60-U dose inhalation of TI Inhalation Powder. Cohort 2 bronchoscopies will occur at 4 hours and again at 8 hours after TI Inhalation Powder. The need to run and the timepoints for bronchoscopies for Cohort 3 will be determined based on the results from Cohort 1 and 2. All subjects will undergo 2 bronchoscopies at Visit 2.

SUMMARY:
Lavage fluid (BAL) is inserted into a lung lobe using a flexible bronchoscope. The fluid is aspirated out to remove any remaining TI. It's performed twice at specific time points in 12 healthy volunteers. BAL fluid will be analyzed for insulin and FDKP.

DETAILED DESCRIPTION:
Informed consent and eligibility occur at Screening. Dosing is at Visit 2. Blood glucose levels are monitored and adjusted using IV infusion of glucose. Bronchoalveolar lavage (BAL) is performed at 30 minutes and 6 hours for Cohort 1 and at 4 and 8 hours for Cohort 2, post TI dose. A series of blood samples are taken at specified timepoints. Cohort 3 will proceed with dosing if deemed necessary once analysis of BAL from Cohorts 1 & 2 is performed. Visit 3 is the follow-up safety visit.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers for greater than or equal to 12 months
* Normal chest x-ray (CXR) at Screening/Visit 1
* Prebronchodilator FEV1 greater than or equal to 80% Third National Health and Nutrition Examination Survey (NHANES) III Predicted
* Prebronchodilator FEV1/FVC greater than or equal to LLN% NHANES III Predicted
* Prebronchodilator total lung capacity (TLC) greater than or equal to 80% of Predicted Intermountain Thoracic Society (ITS)
* Prebronchodilator Dlco (unc) greater than or equal to 80% Predicted (Miller)
* Written Informed Consent

Exclusion Criteria:

* History of diabetes mellitus
* Previous exposure to TI Inhalation Powder within 3 months of Visit 1, or exposure to any other inhaled insulin product
* Allergy or known hypersensitivity to insulin or to any of the drugs to be used in the trial or a history of hypersensitivity to TI Inhalation Powder or to drugs with a similar chemical structure.
* History of chronic obstructive pulmonary disease (COPD), asthma, and or any other clinically important pulmonary disease (eg, cystic fibrosis, bronchiectasis, and/or sleep apnea) confirmed by PFTs and/or radiologic findings.
* Known allergic or adverse reactions to specified medications
* Seizure disorder, significant cardiovascular dysfunction and/or history within 3 months of Visit 1, uncontrolled hypertension, known history of aortic or cerebral aneurysm, renal dysfunction or disease, serum creatinine > 2.0 mg/dL in males and > 1.8 mg/dL in females and/or blood urea nitrogen (BUN) > 50 mg/dL
* Cancer (other than excised cutaneous basal cell carcinoma) within the past 5 years or any history of lung neoplasms.
* History of active viral and/or cirrhotic hepatic disease and/or abnormal liver enzymes, as evidenced by serum aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT) ? 3x upper limit of normal (ULN).
* Active infection (eg, human immunodeficiency virus (HIV), hepatitis) or history of severe infection within 30 days of Visit 1
* Anemia (hemoglobin value ? 10.5 g/dL for females or ? 11.5 g/dL for males.
* Diagnosis of systemic autoimmune or collagen vascular disease requiring previous or current treatment with systemic corticosteroids, cytotoxic drugs, or penicillamine.
* Current or previous chemotherapy, radiation therapy, or amiodarone use that may result in pulmonary toxicity.
* Clinically significant abnormalities or screening laboratory evaluation (unless approved by the Medical Monitor).
* Female subjects who are pregnant, lactating, or planning to become pregnant during the clinical trial period.
* Female subjects of childbearing potential not practicing adequate birth control.
* Current drug or alcohol abuse or a history of drug or alcohol abuse, that, in the opinion of the PI, would not make the subject a suitable candidate for participation in the clinical trial.
* Exposure to any investigational medications or devices within the previous 30 days prior to trial entry or participation in another clinical trial while participating in the clinical trial.
* Unable and/or unlikely to comprehend and/or follow the trial protocol.
* Unable and/or unlikely to comprehend how to use the MedTone Inhaler Model D or inability to properly use the device.
* A lack of compliance with medication or procedures, that, in the PI's opinion, may affect the clinical trial data or the subject's safety and which precludes the subject from further participation in the clinical trial
* Any other concurrent medical or major psychiatric condition that, in the opinion of the PI, makes the subject unsuitable for the clinical trial, or could limit the validity of the informed consent, and/or impair the subject's ability to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Estimation of the amount of insulin in the lungs and amount of FDKP by analyzing BAL fluid, obtained by a flexible fiber optic bronchoscope at various time points after admin of TI Inhalation Powder. | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boss, MD, MPH, Study Chair — Mannkind Corporation
Locations (1):
- PACT Pulmonary Associates, Phoenix, Arizona, United States